CLINICAL TRIAL: NCT05262023
Title: A Phase 1/2, Multicenter, Randomized, Placebo-Controlled, Double Blind Single Dose and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL593 in Healthy Participants and Participants With Frontotemporal Dementia Followed by an Open-Label Extension
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL593 in Healthy Participants and Participants With Frontotemporal Dementia (FTD-GRN)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-H-0001; 2023-508697-28-00 (EU CTIS Number); 2021-005733-16 (EudraCT Number)
Record Dates: First submitted 2022-02-01; First posted 2022-03-02 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Frontotemporal Dementia
Keywords: FTD; FTD-GRN; granulin
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- DNL593 (Healthy Participant) (Experimental)
  Interventions: Drug: DNL593
- Placebo (Healthy Participant) (Placebo Comparator)
  Interventions: Drug: Placebo
- DNL593 (Participants with FTD) (Experimental)
  Interventions: Drug: DNL593
- Placebo (Participants with FTD) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNL593 — Ascending single doses (for healthy participants) and multiple doses (for participants with FTD)
  Arms: DNL593 (Healthy Participant); DNL593 (Participants with FTD)
Drug: Placebo — Ascending single doses (for healthy participants) and multiple doses (for participants with FTD)
  Arms: Placebo (Healthy Participant); Placebo (Participants with FTD)

SUMMARY:
This is a Phase 1/2, multicenter, randomized, placebo-controlled, double-blind study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single and multiple doses of DNL593 in two parts followed by an optional open-label extension (OLE) period.

Part A will evaluate the safety, tolerability, PK, and PD of single doses of DNL593 in healthy male and healthy female participants of nonchildbearing potential. Part B will evaluate the safety, tolerability, PK, and PD of multiple doses of DNL593 in participants with frontotemporal dementia (FTD) over 25 weeks. Part B will be followed by Part C, an optional 18-month OLE period available for all participants who complete Part B.

ELIGIBILITY:
Key Inclusion Criteria:

Part A:

* Women of non-childbearing potential (surgically sterilized or post menopausal) or men, aged ≥18 to ≤ 55 years
* BMI of ≥ 18 to ≤ 32 kg/m²
* When engaging in sex with a woman of child bearing potential, two forms of birth control are required

Part B:

* Women of non-childbearing potential (surgically sterilized or post menopausal) or men, aged ≥18 to ≤ 80 years. Women who are of childbearing potential but on highly effective, low user dependent contraceptive methods will be allowed.
* BMI of ≥ 18 to ≤ 32 kg/m²
* Have a Clinical Dementia Rating® plus National Alzheimer's Coordinating Center frontotemporal lobar degeneration global score ≥ 0.5
* Have confirmed granulin (GRN) mutation via genetic testing or historical records available for review by investigator
* When engaging in sex with a woman of child bearing potential, both the male participant and his female partner must use highly effective contraception

Part C:

* All participants who completed Part B of this trial are eligible for an 18-month OLE if the participant has no unresolved clinically significant TEAEs, where continued dosing may represent a risk to participant safety.

Key Exclusion Criteria:

* Have any history of clinically significant neurologic, psychiatric, endocrine, pulmonary, cardiovascular, gastrointestinal, hepatic, pancreatic, renal, metabolic, hematologic, immunologic, or allergic disease, or other major disorders
* Have a history of malignancy, except fully resected basal cell carcinoma or other malignancies at low risk of recurrence
* Have a clinically significant history of stroke, cognitive impairment due to causes other than FTD, seizure within 5 years of screening, or head trauma with loss of consciousness within 2 years of screening
* Have a positive serum pregnancy test or are currently lactating or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and seriousness of treatment-emergent adverse events (TEAEs) | up to 18 months
Incidence of treatment-emergent clinically significant abnormalities in safety laboratory values | up to 18 months
Change from baseline in vital sign measurements: systolic and diastolic blood pressure | up to 18 months
Change from baseline in vital sign measurements: heart rate | up to 18 months
Change from baseline in vital sign measurements: respiratory rate | up to 18 months
Change from baseline in vital sign measurements: body temperature | up to 18 months
Change from baseline in electrocardiogram (ECG) results including PR, QRS, and QTcF intervals | up to 18 months
Incidence of treatment-emergent clinically significant abnormalities in physical/neurological examination findings | up to 18 months
Change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS; Parts B and C only) | up to 18 months

SECONDARY OUTCOMES:
PK Parameter: Maximum concentration (Cmax) of DNL593 in serum | up to 18 months
PK Parameter: Time to reach maximum concentration (tmax) of DNL593 in serum | up to 18 months
PK Parameter: Area under the concentration-time curve (AUC) from time zero to time of last measurable concentration (AUClast) of DNL593 in serum | up to 18 months
PK Parameter: terminal elimination half-life (t1/2) of DNL593 in serum | up to 18 months
PK Parameter: AUC from time zero to infinity (AUC∞) of DNL593 in serum (Part A only) | up to 84 days
PK Parameter: Accumulation ratio of DNL593 in serum (Parts B and C only) | up to 18 months
PK Parameter: Trough concentration of DNL593 in serum (Ctrough) (Parts B and C only) | up to 18 months
PK Parameter: AUC from time 0 to the end of the dosing interval (AUCτ) of DNL593 in serum (Parts B and C only) | up to 18 months
Concentration of DNL593 in cerebrospinal fluid (CSF) | up to 18 months
DNL593 CSF:serum concentration ratio | up to 18 months
Percentage change from baseline in plasma NfL | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy Berger, MD, Study Director — Denali Therapeutics Inc.
Locations (26):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - John Hopkins University, Baltimore, Maryland
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- Belgium (2):
  - University of Antwerp, Antwerp
  - UZ Leuven, Leuven
- Brazil (2):
  - L2IP - Instituto de Pesquisas Clinicas LTDA, Brasília
  - Faculdade de Medicina Da Universidade de São Paulo, São Paulo
- Colombia (2):
  - Hospital Universitario San Ignacio, Bogotá
  - Grupo de Neurosicencias de la Universidad de Antioquia, Medellín
- Fakultni nemocnice v Motole, Prague, Czechia
- France (3):
  - CHU de Nantes, Nantes
  - CHU Rouen, Rouen
  - CHU Toulouse, Toulouse
- Italy (4):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Istituto Auxologico Italiano, Milan
  - Azienda Ospedaliera Cardinale G Panico, Tricase
- Erasmus University Medical Center, Rotterdam, Netherlands
- Portugal (2):
  - Hospital de Braga, Braga
  - Campus Neurológico Sénior, Torres Vedras
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Guipúzcoa
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
- Turkey (Türkiye) (2):
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Ondokuz Mayis University Hospital, Samsun
- Simbec Orion, Merthyr Tydfil, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No